CLINICAL TRIAL: NCT02316054
Title: Long-term Additive Prognostic Value of Heterogeneity Myocardial Perfusion Imaging of SPECT Over Clinical and Ischemia in High-risk Diabetic Patients.
Brief Title: Evaluation of Myocardial Perfusion Heterogeneity Imaging in Diabetes Patients (EVADIAB)
Acronym: EVADIAB
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-02
Record Dates: First submitted 2014-12-02; First posted 2014-12-12 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes mellitus; coronary microvascular disease; coronary artery disease; myocardial perfusion imaging; prognosis; atherosclerosis; myocardial ischemia; coronary heart disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Microvascular Angina; Coronary Artery Disease; Atherosclerosis; Myocardial Ischemia; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- diabetes and MPHI: myocardial perfusion heterogeneity imaging
  Interventions: Device: MPHI

INTERVENTIONS:
Device: MPHI — addictive value of MPHI to management of high risk cardiovascular type 2 diabetes

SUMMARY:
Long-term additive prognostic value of heterogeneity myocardial perfusion imaging of SPECT over clinical and ischemia in high-risk diabetic patients

DETAILED DESCRIPTION:
Currently, type II diabetes mellitus (DM), has reached epidemic levels in the world. Risk stratification is paramount in patients with DM due to not all patients with DM have a similar cardiovascular (CV) risk. Imaging has thus taken a central role in the assessment of CV health and in the diagnosis, evaluation, and management of CV diseases in DM. The prognostic value of relative myocardial perfusion imaging (MPI) using single-photon emission tomography (SPECT) is well established. Consistent with this data, DM patients with abnormal relative MPI results also have higher rates of death and non-fatal MI than those with normal results. However, DM patients with normal stress tests also have higher rates of cardiac events than non-DM counterparts with normal tests and despite that most guidelines recommend a systematic screening of asymptomatic high risk patients with diabetes for silent ischemia, real benefit of this strategy has not been demonstrated compared with optimal medical treatment without ischemia detection. New more sensitive noninvasive imaging to assess MPI abnormalities is needed.

Coronary microvascular dysfunction (CMVD) is closely associated with coronary artery disease; it is an independent risk factor and predicts future coronary events or clinically manifest disease up to 10 years later. To date, non-invasive measurement of CMVD myocardial perfusion heterogeneity imaging (MPHI) by SPECT is not available into clinical practice. We developed a new method to study the CMVD by SPECT. In this study, we use a mathematic technique from entropy analysis to provide precise, objective, automated quantification of MPHI at stress and at rest with SPECT. We sought to assess the prognostic value of MPHI in high-risk diabetic patients being investigated for ischemia. Therefore, we prospectively evaluated the incremental prognostic value of MPHI in patients with type 2 DM during long-term follow-up. Coronary microvascular dysfunction is closely associated with coronary artery disease; it is an independent risk factor and predicts future coronary events or clinically manifest disease up to 10 years later.

In this study, we use a new mathematic technique from entropy analysis to provide precise, objective, automated quantification of perfusion heterogeneity at stress with camera SPECT. This method may be a non-invasive imaging to assess coronary microvascular dysfunction.

The main hypothesis is that the presence of myocardial perfusion heterogeneity is predictive of 5-year cardiovascular events in patients referred to the Nuclear Cardiology Department for routine evaluation of known or suspected CAD in diabetes patients with very high risk cardiovascular.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Clinical indication for myocardial perfusion imaging
* Diabetics with very high risk of cardiovascular events defined by the SCORE risk

Exclusion Criteria:

* Pregnant woman
* Breast feeding women
* Severe comorbidity with life expectancy 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: high-risk cardiovascular type 2 diabetic patients
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2007-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
cardiac death,or Q-wave myocardial infarction (MI), or the need for myocardial revascularization > 3 months after SPECT | 4 years
  Composite outcome: cardiac death, Q-wave myocardial infarction (MI), the need for myocardial revascularization > 3 months after SPECT

SECONDARY OUTCOMES:
cardiac death | 4 years
  death from coronary artery disease, heart failure or sudden death
non fatal myocardial infarction | 4 years
  non fatal myocardial infarction
myocardial revascularization > 3 months after SPECT | 2 years
  myocardial revascularization > 3 months after SPECT

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Barone-Rochette, MD,PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- university Hospital, Grenoble, France

REFERENCES:
- [Derived] Djaileb L, Seiller A, Canu M, De Leiris N, Martin A, Poujol J, Fraguas-Rubio A, Leenhardt J, Carabelli A, Calizzano A, De Fondaumiere M, Broisat A, Desvignes M, Vanzetto G, Ghezzi C, Fagret D, Riou LM, Barone-Rochette G. Prognostic value of SPECT myocardial perfusion entropy in high-risk type 2 diabetic patients. Eur J Nucl Med Mol Imaging. 2021 Jun;48(6):1813-1821. doi: 10.1007/s00259-020-05110-4. Epub 2020 Nov 20. PMID 33219463